CLINICAL TRIAL: NCT03481452
Title: NBO Ameliorates Disorders of Regulation of States in Little Infants From Perinatal Anxiety
Brief Title: Tutorial of Clinical Trial Registration
Acronym: CTREG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: Xian Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU-PRENATALSTRESS-001; XCH-PRENATALSTRESS-001 (Other: Xi'an Children's Hospital)
Record Dates: First submitted 2017-11-30; First posted 2018-03-29 (Actual); Last update posted 2018-04-03 (Actual); Status verified 2018-01

CONDITIONS: Behavior; Anxiety
Keywords: anxiety; regulation of states; NBO; HAMA
MeSH Terms: conditions — Behavior; Anxiety Disorders | interventions — Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- psychotherapy intervention group (Experimental): NBO behavioral intervention would be used to improve mother-infant dyad interaction and infants' disorders of regulation of states.
  Interventions: Behavioral: psychotherapy
- control group (No Intervention): No behavioral intervention would be used.

INTERVENTIONS:
Behavioral: psychotherapy — NBO is an infant-focused, family relationship-based intervention measure, which aims to exhibit to parents infants' surprised ability, understand infants' strength and aspects needed to be improved, strength parents' parenting confidence, and promote sound development of infant-mother relationship.
  Other Names: Neonatal Behavioral Observation (NBO)
  Arms: psychotherapy intervention group

SUMMARY:
The present study aimed to determine whether infants disorders of regulation of states are associated with perinatal anxiety, and further to explore the efficacy of the behavioral intervention in enhancing positive interactions between mothers and their infants and thus ameliorating infants' disorders of regulation of states.

DETAILED DESCRIPTION:
The subjects were recruited from the hospitalized pregnant women waiting for delivery from the department of gynecology and obstetrics of the first affiliated hospital of Xi'an Jiaotong university. A total of 200 perinatal anxiety women were divided to two group(behavioral intervention group and control group) according to mental health assessment. Inclusion criteria were applied: 1. mother aged 18-40 years; 2. First-time mother, full-term and singleton pregnancy; 3.the Hamilton Anxiety Scale(HAMA) score ≥14; 4.birth with no intrapartum complications; and 5. Apgar score > 8 at the first, fifth, and tenth minutes after birth. Exclusion criteria were as follows: any mental illness besides anxiety, maternal medical illness, hypertension, advanced liver disease, renal failure, cancer, valvular heart disease, heart failure, stroke,atrial fibrillation, peripheral arterial disease, and other severe diseases.Preterm infants (< 37 weeks gestation) and multiple births were excluded from the current analysis. All the subjects completed the infants behavior and regulation of states assessment by the NBAS and were followed to 8 weeks postpartum. Mother-newborn pairs were randomly divided into NBO intervention group and control group. NBO intervention was performed once a week until 2 months. 2 ml peripheral blood was collected in the pregnant woman before delivery and in the newborns within 3 days postpartum.The serum fraction was removed after centrifugation and stored at -20°C. Levels of serum cortisol in mothers and newborns were determined using Chemiluminescence analysis (CLIA) and a radio immunoassay. All sample analyses were performed by the first affiliated hospital of Xi'an Jiaotong university chemistry laboratory. Laboratory personnel were blinded to mother and infant outcomes.

ELIGIBILITY:
Inclusion Criteria:

* mother aged 18-40 years;
* first-time mother, full-term and singleton pregnancy;
* the Hamilton Anxiety Scale(HAMA) score ≥14;
* the birth with no intrapartum complications;
* Apgar score > 8 at the first, fifth, and tenth minutes after birth.

Exclusion Criteria:

* any mental illness besides anxiety, maternal medical illness, hypertension, advanced liver disease, renal failure, cancer, valvular heart disease, heart failure, stroke, atrial fibrillation, peripheral arterial disease, and other severe diseases;
* preterm infants (< 37 weeks gestation);
* multiple births;
* infants with congenital anomalies, signs of illness, or high-risk factors.

Max Age: 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
NBO ameliorates disorders of regulation of states in little infants from perinatal anxiety | up to 2 months
  The Hamilton Anxiety Scale(HAMA) was used to assess mothers anxiety state and whose score ≥14 were included. Meanwhile, Neonatal Behavioral Assessment Scale (NBAS) was used to assess infants neurobehavioral development and regulation of states from birth to 2 months. Regulation of states in the NBAS including four parts: cuddliness、consolability 、self-quieting and hand-to-mouth. Every part scores from 1 to 9, and the 1 represents worst and 9 for best. Higher scores of NBAS is associated with better regulation of states. Newborn Behavioral Observations (NBO) would be used to improve mother-infant dyad interaction and ameliorates infants disorders of regulation of states. Mother-newborn pairs were randomly divided into NBO intervention group and control group. NBO intervention was performed once a week until 2 months. Mother-newborn pairs serum would be collected to measure cortisol.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Li, PhD, MD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Undecided